CLINICAL TRIAL: NCT03548870
Title: Effects of Transcutaneous Electrical Nerve Stimulation During Acute Aerobic Exercise in Patients With Chronic Obstructive Pulmonary Disease After Exacerbation
Brief Title: Transcutaneous Electrical Nerve Stimulation During Exercise in Patients With COPD
Acronym: proTENS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough recruitment
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-A02290-53
Record Dates: First submitted 2018-05-17; First posted 2018-06-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD; Physical Activity; Rehabilitation; TEN
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: sham transcutaneous electrical nerve stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test with TENS (Experimental): Patients will perform one Constant Work-Rate Exercise Test at 80% of maximum workload with low frequency TENS
  Interventions: Other: CWRT with low frequency transcutaneous electrical nerve stimulation
- Test with sham-TENS (Sham Comparator): Patients will perform one Constant Work-Rate Exercise Test at 80% of maximum workload with low frequency sham-TENS
  Interventions: Other: CWRT with sham-low frequency transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: CWRT with low frequency transcutaneous electrical nerve stimulation — 4 self adhesive surface electrodes will be positioned by pair on quadriceps. Patients will have a low frequency TENS for 20 min at rest. During this period, intensity will be increased every 5 minutes to the maximum tolerated by the patient (below pain threshold, sensation strong but comfortable). Thereafter, intensity is not increased anymore during the test.
  Current characteristics : Rehab 400, CefarCompex 5Hz 200 µs frequency bidirectional
  Arms: Test with TENS
Other: CWRT with sham-low frequency transcutaneous electrical nerve stimulation — 4 self adhesive surface electrodes are positioned by pair on quadriceps. Patients will have a sham-low frequency TENS for 20 min at rest. During this period, intensity will be increased for 1 minute to the maximum tolerated by the patient. After this procedure, intensity will be progressively setted back to 1mA. Current characteristics : Rehab 400, CefarCompex 5Hz 200 µs frequency bidirectional
  Arms: Test with sham-TENS

SUMMARY:
Early pulmonary rehabilitation is recommended after an episode of severe exacerbation of chronic obstructive pulmonary disease (COPD). However, its implementation is challenging particularly as regard exercise training. Several studies showed that transcutaneous electrical nerve stimulation (TENS) could improve dyspnea and pulmonary function. The aim of this study is to assess the acute effect of TENS on exercise tolerance in post-exacerbation COPD patients

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD

Exclusion Criteria:

* exercise contraindication Any musculoskeletal problems, cardiovascular or
* neurological comorbidities that limits exercise.
* pH < 7,35
* Body temperature > 38°C
* cardiac frequency > 100 bpm at rest
* systolic blood pressure < 100 mmHg
* exacerbation during the study
* heart pace-maker or defibrillator
* Opiate treatment during the last 3 months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
comparison of exercise tolerance | two CWRET will be carried out in different days, separate from 24 hours minimum for a total time frame of 5 days maximum
  Comparison of endurance time (Tlim, in second) during constant workload testing (CWRET) under 2 conditions

SECONDARY OUTCOMES:
Difference in peripheral muscle oxygenation | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Muscle oxygenation (arbitrary unit) will be evaluated using Near-infrared spectroscopy technology.
Difference in Dyspnea | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in dyspnea using Modified Borg Scale (0 - 10 points) 0=no dyspnea ; 10 = maximal effort
Difference in Oxygen Saturation | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in Oxygen Saturation (%) using a pulse oximetry (SpO2)
Difference in Cardiac Frequency | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in Cardiac Frequence (bpm) using a pulse oximetry
Difference in muscular fatigue | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in muscular fatigue using Modified Borg Scale (0 - 10 points) 0=no muscular fatigue ; 10 = maximal effort
Difference in oxygen consumption | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in oxygen consumption (milliliters per minute) will be measured breath-by-breath using a computer-based exercise system
Difference in carbon dioxide production | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in carbon dioxide production (milliliters per minute) will be measured breath-by-breath using a computer-based exercise system
Difference in minute ventilation | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in minute ventilation (liters per minute) will be measured breath-by-breath using a computer-based exercise system
Difference in tidal volume | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in tidal volume (Liters) will be measured breath-by-breath using a computer-based exercise system
Difference in respiratory rate | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in respiratory rate (cycles per minute) will be measured breath-by-breath using a computer-based exercise system
Difference in inspiratory capacity | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in inspiratory capacity (Liters) will be measured breath-by-breath using a computer-based exercise system
Difference in respiratory quotient | The outcome will be measure during every CWRET. The two CWRET will be carried out in different days, separate from 24H minimum for a total time frame of 5 days maximum. Data will be continuously collected during exercise
  Difference in respiratory quotient (ratio) will be measured breath-by-breath using a computer-based exercise system

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier du Havre, Montivilliers, France

IPD SHARING:
Plan to Share IPD: Undecided